CLINICAL TRIAL: NCT01726179
Title: Efficacy of Resin Infiltration of Proximal Caries Lesions in Primary Molars: Randomized Clinical Trial
Brief Title: Efficacy of Proximal Caries Infiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Collaborators: Universidade Federal do Rio de Janeiro (Other); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECIPRJ13
Record Dates: First submitted 2012-11-01; First posted 2012-11-14 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Dental Health; Caries
Keywords: caries infiltration; caries arrest; dental anxiety; dental stress; resin infiltration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resin infiltration (Experimental): This study is a split mouth design. One tooth with a proximal caries lesion is randomized into this arm and another tooth to the arm "Control". Teeth in this arm are treated by the resin infiltration technique using Icon (DMG, Germany) according to manufactures´ instructions. In addition patients and their guardians are instructed to floss once a day and to brush with fluoridated toothpaste twice a day.
  Digital bitewing radiographs will be taken at baseline and repeated after 12 months. Additionally caries risk will be evaluated.
  Interventions: Device: Resin infiltration
- Control (Other): This study is a split mouth design. One tooth with a proximal caries lesion is randomized into this arm and another tooth to the arm "Resin infiltration". Teeth randomized into this arm do not recieve any special treatment except general oral nonivasiv treatment (flossing and brushing). Patients and their guardians are instructed to floss once a day and to brush with fluoridated toothpaste twice a day.
  Digital bitewing radiographs will be taken at baseline and repeated after 12 months. Additionally caries risk will be evaluated.
  Interventions: Device: Control

INTERVENTIONS:
Device: Resin infiltration — Proximal caries lesions that are selected for this intervention will be treated with the resin infiltrant Icon according to the manufacturer's instructions. In short, local anesthesia of the gingival papila, application of rubber dam, etching of the lesion surface for 120 s using 15%HCl gel, washing the lesion with water spray for 30 s, drying the lesion with 100% ethanol for 30 s and subsequent air blowing, application of the infiltrant for 180 s using an applicator provided with the kit, removing excess material from the lesion surface by air blowing and flossing, light curing of the infiltrant for 40 s, repeated application for 60 s, light curing for 40 s, polishing, and removal of the rubber dam.
  Other Names: Icon (DMG, Germany), Approximal resin infiltration kit
  Arms: Resin infiltration
Device: Control — Proximal caries lesions do not recieve a placebo treatment, but simply left untreated.
  Arms: Control

SUMMARY:
The goal of the project is to investigate the clinical efficacy of management of early caries lesions by resin infiltration and to further scrutinize the patient stress experiences.

DETAILED DESCRIPTION:
The aim of this study is to test the clinical efficacy of caries infiltration to arrest proximal caries lesions in primary molars. It was hypothesized that infiltrated lesions (test lesions) will progress significantly less than non infiltrated lesions (control lesions). Additionally, it was hypothesized that dental anxiety and stress related to caries infiltration will be significantly less than dental anxiety related to a conventional restorative procedure. The study will be a controlled clinical trial with a split mouth design and blind evaluation of the outcome (caries progression). Caries progression will be evaluated annually, 12, 24, and 36 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* children with one tooth surface with active caries lesions
* two primary molars with proximal lesion detected on the x-ray (scores 2 (E2) or 3 (D1) in Mejàre et al. scoring system with less depth
* asigned informed consent.

Exclusion Criteria:

* children who do not cooperate during dental appointments
* primary molars supposed to exfoliate in less than two years
* lesions showing obvious cavitation or clear sings of inactivity

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Caries progression rate | 1 year
  Radiographic evaluation of infiltrated and control caries lesions to evaluate caries progression. This is done by pairwise comparison of digital bitewing radiographs by one calibrated, blinded examiner.

SECONDARY OUTCOMES:
Stress reaction during treatment | Immediate
  To evaluate dental anxiety and stress reactions in relation to the caries infiltration procedure in comparison with a dental examination appointment and conventional resin restoration appointment.
  A facial image scale with five faces ranging from very happy (1) to very unhappy (5) will be used.
Caries risk | Baseline, 6 months, 1 year, 2 years, 3 years
  Caries risk is asses based on caries index (Nyvad criteria), proximal plaque index (0 = no visible plaque; 1 = visible plaque) and gingival bleeding index (0 = no bleeding after flossing; 1 = bleeding after flossing), dietary habits, and exposition to fluorides based on the Cariogram model.
Caries progression rate | 2 years, 3 years
  Radiographic evaluation of infiltrated and control caries lesions to evaluate caries progression in long term. This is done by pairwise comparison of digital bitewing radiographs by one calibrated, blinded examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Vera M Soviero, Prof., Dr., Principal Investigator — Universidade do Estado do Rio de Janeiro, Faculdade de Odontologia
Locations (1):
- Universidade do Estado do Rio de Janeiro, Faculdade de Odontologia., Rio de Janeiro, Brazil

REFERENCES:
- [Result] Ammari MM, Jorge RC, Souza IPR, Soviero VM. Efficacy of resin infiltration of proximal caries in primary molars: 1-year follow-up of a split-mouth randomized controlled clinical trial. Clin Oral Investig. 2018 Apr;22(3):1355-1362. doi: 10.1007/s00784-017-2227-7. Epub 2017 Oct 8. PMID 28990122
- [Result] Jorge RC, Ammari MM, Soviero VM, Souza IPR. Randomized controlled clinical trial of resin infiltration in primary molars: 2 years follow-up. J Dent. 2019 Nov;90:103184. doi: 10.1016/j.jdent.2019.103184. Epub 2019 Aug 26. PMID 31465818